CLINICAL TRIAL: NCT00257322
Title: A Pilot Study of Cellular Immune Augmentation in Colon and Rectal Cancer Therapy
Brief Title: Cellular Immune Augmentation in Colon and Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Chao Family Comprehensive Cancer Center, Cancer Center, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 02-60; 2003-2876 (Other: University of California, Irvine)
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Results first posted 2016-04-26 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-02

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: Metastatic colon cancer; Metastatic rectal cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GM-CSF (Experimental): Granulocyte-macrophage colony-stimulating factor (GM-CSF) 250ug/m^2 SQ QD with a cap of 500mcg SQ QD
  Interventions: Drug: GM-CSF

INTERVENTIONS:
Drug: GM-CSF — 250ug/m^2 SQ QD with a cap of 500mcg SQ QD

SUMMARY:
While new treatments for metastatic and recurrent colorectal cancer have become available over the past several years, this disease remains incurable with a limited life expectancy from the time of diagnosis. New strategies for treatment of disseminated colorectal cancer are needed. Under this proposal, patients with advanced colorectal cancer will receive Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) to stimulate endogenous dendritic cells and enhance anti-tumor immune mechanisms. This will be combined with standard chemotherapy and patients will be followed for response and overall survival. Detailed correlative laboratory analysis will also be performed to define the extent of dendritic cell and cellular immune system stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have: metastatic, disseminated or recurrent colon or rectal cancer
* Patient to receive weekly or biweekly chemotherapy for at least 4 cycles (4 weeks) Examples include: 5FU or 5FU/leucovorin given once weekly Irinotecan (single agent) given once weekly 5FU/leucovorin/irinotecan given once weekly
* Patient must be able to be taught to administer GM-CSF subcutaneously

Exclusion criteria:

* Known allergic or other adverse reaction to GM-CSF
* Chemotherapy administration more frequently than bi-weekly
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-04; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall Holcombe, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinez M, Ono N, Planutiene M, Planutis K, Nelson EL, Holcombe RF. Granulocyte-macrophage stimulating factor (GM-CSF) increases circulating dendritic cells but does not abrogate suppression of adaptive cellular immunity in patients with metastatic colorectal cancer receiving chemotherapy. Cancer Cell Int. 2012 Jan 23;12(1):2. doi: 10.1186/1475-2867-12-2. PMID 22270330

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 subjects enrolled between Jun 2003 and Jan 2007 in UCIMC location. All subjects undergoing treatment are presented with all options for their care - research or non-research.
Pre-assignment Details: Subjects with known allergic or other adverse reaction to GM-CSF are excluded from study. Also pregnant and lactating women were excluded from study.
Groups:
- Chemo Therapy and GM-CSF: Granulocyte-macrophage colony-stimulating factor (GM-CSF) 250ug/m^2 SQ QD with a cap of 500mcg SQ QD
Period: Overall Study
Arm/Group | Chemo Therapy and GM-CSF
Started | 20 (20 subjects accrued.)
Completed | 16 (4 subjects withdrew from this study.)
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Chemo Therapy and GM-CSF: Granulocyte-Macrophage Colony-Stimulating Factor
Arm/Group | Chemo Therapy and GM-CSF
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.65 (13.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Secondary Outcome: Response Rates and Overall Survival.
Description: Effect of cellular immune stimulation on response rates and overall survival. This is a secondary endpoint and while data will be recorded, a larger study with improved power will be necessary to confirm any improvements noted.
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Chemo Therapy and GM-CSF
Number analyzed (Participants) | 16
Participants
  Response Rates | 16
  Overall Survival | 16

2. Primary Outcome: Participants Exhibiting Immune Response
Description: Immunological dendritic cell and cellular immune responses to GM-CSF administered in conjunction with chemotherapy for patients with advanced colorectal cancer.
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Chemo Therapy and GM-CSF
Number analyzed (Participants) | 16
Participants | 11

ADVERSE EVENTS:
Arm/Group | Chemo Therapy and GM-CSF
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No